CLINICAL TRIAL: NCT05326113
Title: Effect of Physiotherapy on the Usage of Proton Pump Inhibitors and Changes in the Pressure of the Lower Esophageal Sphincter in Patients With Achalasia After Per Oral Endoscopic Myotomy
Brief Title: The Effect of Physiotherapy on Post POEM Reflux
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Doc. (Ass. prof.) Jan Martinek, MD, PhD, AGAF, Prof., Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IClinicalEM4
Record Dates: First submitted 2022-03-15; First posted 2022-04-13 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Reflux, Gastroesophageal; Achalasia; Esophagitis
Keywords: Per-oral endoscopic myotomy; Reflux; Physiotherapy; Proton pump inhibitors; Diapraghm; Achalasia; Lower esophageal sphincter
MeSH Terms: conditions — Gastroesophageal Reflux; Esophageal Achalasia; Esophagitis | interventions — Physical Therapy Modalities; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy (Experimental): Patients will undergo physiotherapy and will be regularly examined by an assigned physician.
  Initial physiotherapy will last 60minutes, other therapies will last 30minutes. Physiotherapy will aim on diaphragmatic breathing and dynamic neuromuscular stabilization exercises. In the 1st month, the patient attends physiotherapy once a week In the 2nd, 3rd and 4th month, the patient attends physiotherapy once every 14 days.
  Symptomatic patients will take PPIs based on the recommendation of the treating physician who will recommend a dose of PPIs. Used PPIs will be Emanera 1x40mg (standard dose), 2x40mg (higher dose) or 1x40mg on demand.
  During the follow-up period, patients may, in agreement with the attending physician, reduce the dose of PPIs (from twice a day to once a day, from once a day to an "on-demand" regime or discontinue them altogether).
  The use of PPIs will be accurately documented.
  Interventions: Other: Physiotherapy
- Control group (Active Comparator): Control group will undergo standard treatment of reflux with PPIs and will be regularly examined by an assigned physician.
  Symptomatic patients will take PPIs based on the recommendation of the treating physician who will recommend a dose of PPIs. Used PPIs will be Emanera 1x40mg (standard dose), 2x40mg (higher dose) or 1x40mg on demand.
  All patients with esophagitis LA A/B/C will be treated with IPP-Emanera 1x40mg for at least 6 weeks at the start of the study.
  During the follow-up period, patients may, in agreement with the attending physician, reduce the dose of PPIs (from twice a day to once a day, from once a day to an "on-demand" regime or discontinue them altogether).
  The use of PPIs will be accurately documented.
  Interventions: Drug: Control group

INTERVENTIONS:
Other: Physiotherapy — After POEM, patient underwent physiotherapy consisting of diaphragmatic breathing and dynamic stabilization exercises and PPIs
  Arms: Physiotherapy
Drug: Control group — All patients will be treated with standard course of PPIs after POEM without physiotherapy.
  Arms: Control group

SUMMARY:
Per-oral endoscopic myotomy has been used as a treatment method of esophageal achalasia. Patients who undergo POEM as a treatment of achalasia are often presented with development of reflux as a side effect of the surgery. Patients are then in need to use proton pump inhibitor drugs as a long term treatment of the reflux symptoms.

Physiotherapy aimed on the strengthening of diaphragm and lower esophageal region is effective in gastroesophageal reflux disease. Therefore we are expecting positive effect of physiotherapy in post POEM patients with reflux symptoms and the possible reduction of PPI drug usage need.

The aim of the study is to objectify the effect of physiotherapy, to describe in detail the used physiotherapeutic techniques and to develop practical guidelines for the treatment of patients after POEM with GERD.

DETAILED DESCRIPTION:
The goal per-oral endoscopic myotomy (POEM) is to release a non-relaxing, often spastic lower esophageal sphincter (LES). During POEM an incision of the esophageal muscle layer (m.propria) is performed using the submucosal tunnel technique.

A complication of POEM is the development of reflux, which occurs in up to 50% of patients (within 12 months), with the occurrence of severe esophagitis being rare. However, patients are treated with proton pump inhibitors (PPIs) after POEM, either daily or on-demand. As a result, patients after POEM are regularly monitored for the possible development of symptomatic or asymptomatic reflux, which (if left untreated) can lead to the development of complications, including Barrett's esophagus, a known precancerous lesion.

The main reason for reflux in patients after POEM is an insufficient function of the LES, which is formed not only by the smooth muscle of the esophagus, but also by the skeletal muscle- diaphragm, which remains intact during the POEM itself. Together, these two structures form a major component of antireflux barriers. Since the crural part of the diaphragm is a skeletal striated muscle, it is a trainable muscle.

The study will involve 30 patients after POEM with diagnosed reflux. Three months after POEM patients undergo follow-up examinations using high resolution manometry, 24hours pH test for reflux and gastroscopy. Based on the results of the examination in the 3rd month after the POEM, those who meet the inclusion criteria, will be offered to participate in this study. Patients will be asked to fill in the quality of life questionnaire of patients after POEM and the validated questionnaire for patients with reflux disease. Patients will be randomized in 2 groups (15 in both arms, ratio 1:1), one group will undergo 4 months of physiotherapy treatment using PPI on demand, second group will be a control group undergoing standard treatment of reflux symptoms with PPI on demand.

This study will evaluate the effect of standard treatment of post-POEM esophageal reflux compared to the effect of physiotherapy using dynamic neuromuscular stabilization in post-POEM patients with esophageal reflux.

There is currently no study looking at the effect of physiotherapy in post-POEM patients, we believe this could be a beneficial study.

If this study demonstrates that physiotherapy alleviates the symptoms of post-POEM reflux, it could be one of the official methods of treatment for this group of patients and thus significantly increase their quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. esophageal achalasia (or other primary motility disease) treated by per oral endoscopic myotomy (POEM)
2. symptomatic post-POEM reflux and/or esophagitis LA A/B/C (grade by The Los Angeles Classification) present 3 months after POEM surgery
3. positive finding on esophageal 24hours pH Test 3 months after POEM surgery
4. signed informed consent

Exclusion Criteria:

1. reflux symptoms previously to the POEM surgery (except regurgitation)
2. repeated POEM surgery
3. Esophagitis of LA grade D
4. asymptomatic pathologic reflux without signs of esophagitis 3 months post POEM surgery (patient is not indicated to use proton pump inhibitor "PPI" drugs)
5. previous gastric surgery
6. patients undergoing cancer treatment
7. pregnancy
8. known allergy or intolerance of proton pump inhibitor drugs
9. other circumstances preventing participation in the study
10. Inability to obtain informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-31 (Actual); Primary Completion 2024-08-18 (Estimated); Study Completion 2025-01-18 (Estimated)

PRIMARY OUTCOMES:
Comparison of proton pump inhibitor drugs usage in experimental and control group | 9-10 months
  Rate of use of IPP and only Emanera 2x40mg (higher dose), 1X40mg (standard dose), or 1x40 mg in case of problems or completely discontinue IPP

SECONDARY OUTCOMES:
Comparison of diagnostic examinations | 9-10 month
  The secondary outputs will be the results of high resolution manometry examinations, where we monitor changes in pressure in the lower esophageal sphincter area and esophageal motility. The positivity and reflux rate will be demonstrated by 24hours pH testing and evaluated according to the De Meester score. Gastroscopy to evaluate the absence or presence of esophagitis.
Comparison of questionnaires | 9-10 months
  Evaluation of the Quality of life questionnaire of patients after POEM. Evaluation of the validated questionnaire for gastroesophageal reflux disease.

CONTACTS AND LOCATIONS:
Overall Officials: Kateřina Mádle, Principal Investigator — Charles University 2nd faculty of medicine, Prague, Czech Republic; Jan Martínek, Principal Investigator — Department of Hepatogastroenterology, Institute for Clinical and Experimental Medicine, Prague, Czech Republic; Zuzana Vacková, Principal Investigator — Department of Hepatogastroenterology, Institute for Clinical and Experimental Medicine, Prague, Czech Republic; Milan Martínek, Principal Investigator — Charles University Faculty of Physical Education and Sport; Lucie Zdrhová, Principal Investigator — Department of Internal Medicine, Pilsen, Czech Republic; Alena Kobesová, Principal Investigator — Charles University 2nd faculty of medicine, Prague, Czech Republic
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided